CLINICAL TRIAL: NCT00178100
Title: Maintenance Therapies in Late-Life Depression 2 (MTLD-2)
Brief Title: Paroxetine and Interpersonal Psychotherapy for Maintaining Health and Well-being in Elderly Individuals With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH043832-02 (NIH); 971156; DATR A4-GPS
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Unipolar Depression
Keywords: Depression; Elderly; Late Life
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Interpersonal Psychotherapy; Paroxetine

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy
Drug: paroxetine

SUMMARY:
This study will evaluate the effectiveness of paroxetine versus interpersonal psychotherapy and a combination of the two in helping elderly patients with depression remain well and improve quality of their lives.

DETAILED DESCRIPTION:
This is primarily a study of maintenance therapies, not a study of acute therapeutic efficacy, in late-life major depression. The study aims to identify factors that encourage maintenance of treatment gains and to identify which patients need which kinds of treatment to remain well. The following questions are to be addressed:

* Is the probability of recurrence different among the treatment groups?
* What variables may be related to, or predictive of, differences among groups?
* After 1 to 2 years of maintenance therapy, will patients assigned to maintenance combined treatment with both paroxetine and interpersonal psychotherapy remain well at higher rates than patients assigned to paroxetine alone, interpersonal psychotherapy alone, or placebo?
* Will the time to recurrence differ across treatment groups, and what variables may be related to, or predictive of, time to recurrence?

The major study hypothesis is that combined treatment with paroxetine and interpersonal psychotherapy will be superior to either treatment alone (and to placebo) in preventing recurrence of major depressive episodes in patients aged 70 and above.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00000377

http://clinicaltrials.gov/show/NCT00177671

ELIGIBILITY:
Inclusion Criteria:

* Age 69 or older
* meets DSM-IV criteria for current unipolar major depression
* HRSD (17 item) score of 15 or higher
* Folstein Mini Mental Status exam score of 18 or higher

Exclusion Criteria:

* Lifetime diagnosis of any psychotic disorder or bipolar disorder
* alcohol or drug abuse within the past six months
* MATTIS Dementia Rating Score of 120 or less
* Contraindication to SSRI therapy
* Hyponatremia

Min Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 225
Dates: Start 1999-03; Study Completion 2005-08

PRIMARY OUTCOMES:
Combined treatment with paroxetine and interpersonal psychotherapy will be superior to either treatment alone (and to placebo)in preventing recurrence of major depressive episodes in patients aged 70 and above.

SECONDARY OUTCOMES:
Cognitive status: Folstein Mini-Mental Status Exam, MATTIS Dementia Rating Scale, EXIT, and CDR
Quality of Life measures: Quality of Wellbeing Scale, CIDI Health Services Utilization, Older American Resources and Services Activities of Daily Living Scale, Global Assessment Scale, PSQI, SF-36, UKU, and CIRS-G
Social Support: Interpersonal Support Evaluation List, Luben Social Network Scale; and Life Events and Difficulties Schedule
Psychiatric status: SCID, Hamilton Depression Rating Scale, Suicidal History Questionnaire, Antidepressant Treatment History Form, Brief Psychiatric Rating Scale, and anxiety subscale of Brief Symptom Inventory
MRI

CONTACTS AND LOCATIONS:
Overall Officials: Charles F Reynolds III, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Reynolds CF 3rd, Dew MA, Pollock BG, Mulsant BH, Frank E, Miller MD, Houck PR, Mazumdar S, Butters MA, Stack JA, Schlernitzauer MA, Whyte EM, Gildengers A, Karp J, Lenze E, Szanto K, Bensasi S, Kupfer DJ. Maintenance treatment of major depression in old age. N Engl J Med. 2006 Mar 16;354(11):1130-8. doi: 10.1056/NEJMoa052619. PMID 16540613
- [Derived] Carreira K, Miller MD, Frank E, Houck PR, Morse JQ, Dew MA, Butters' MA, Reynolds CF 3rd. A controlled evaluation of monthly maintenance interpersonal psychotherapy in late-life depression with varying levels of cognitive function. Int J Geriatr Psychiatry. 2008 Nov;23(11):1110-3. doi: 10.1002/gps.2031. PMID 18457338